CLINICAL TRIAL: NCT01767155
Title: Randomized Controlled Study Comparing AEZS-108 With Doxorubicin as Second Line Therapy for Locally Advanced, Recurrent or Metastatic Endometrial Cancer.
Brief Title: Zoptarelin Doxorubicin (AEZS 108) as Second Line Therapy for Endometrial Cancer
Acronym: ZoptEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEZS-108-050
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — LHRH, lysine(6)-doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AEZS-108 / zoptarelin doxorubicin (Experimental): 267 mg/m^2 by 2-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles up to 9 cycles
  Interventions: Drug: AEZS-108 / zoptarelin doxorubicin
- doxorubicin/ standard chemotherapy (Active Comparator): 60 mg/m^2 by intravenous bolus injection or 1-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles
  Interventions: Drug: doxorubicin

INTERVENTIONS:
Drug: AEZS-108 / zoptarelin doxorubicin — 267 mg/m^2 by 2-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles for a maximum of 9 cycles
  Other Names: AEZS-108
  Arms: AEZS-108 / zoptarelin doxorubicin
Drug: doxorubicin — 60 mg/m^2 by intravenous bolus injection or 1-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles
  Arms: doxorubicin/ standard chemotherapy

SUMMARY:
Open-label, randomized, active-controlled, two-arm Phase III study to compare the efficacy and safety of AEZS-108 and doxorubicin.

DETAILED DESCRIPTION:
The study will include about 500 patients with endometrial cancer resistant to platinum/taxane-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years of age
2. Histologically confirmed endometrial cancer
3. Advanced (FIGO stage III or IV), recurrent or metastatic disease.
4. Measurable or non-measurable disease that has progressed since last treatment.
5. 5. Patients with advanced, recurrent or metastatic endometrial cancer who have received one chemotherapeutic regimen with platinum and taxane (either as adjuvant or as first line treatment) and who have progressed.
6. Availability of fresh or archival FFPE (formalin-fixed and paraffin-embedded) tumor specimens for analysis of LHRH (luteinizing hormone releasing hormone) receptor expression.

Exclusion Criteria:

1. ECOG (Eastern Cooperative Oncology Group) performance status > 2.
2. Inadequate hematologic, hepatic or renal function
3. Red blood cell transfusion within 2 weeks prior to anticipated start of study treatment.
4. History of myocardial infarction, acute inflammatory heart disease, unstable angina, or uncontrolled arrhythmia within the past 6 months.
5. Impaired cardiac function defined as left ventricular ejection fraction (LVEF) < 50 % (or below the study site's lower limit of normal) as measured by MUGA (multigated radionuclide angiography) or ECHO (echocardiography).
6. Concomitant use of prohibited therapy (specified in protocol)
7. Chemo-, immune-, or hormone-therapy within 5 elimination half life times or 4 weeks prior to randomization, whichever is the shorter. Radiotherapy (including pre- or post-operative brachytherapy) within 4 weeks prior to randomization.
8. Previous anthracycline-based chemotherapy (daunorubicin, doxorubicin, epirubicin, idarubicin, mitoxantrone and valrubicin), in any formulation.
9. Anticipated ongoing concomitant anticancer therapy during the study.
10. History of serious co-morbidity or uncontrolled illness that would preclude study therapy, such as active tuberculosis or any other active infection.
11. Brain metastasis, leptomeningeal disease.
12. Pregnant or lactating female or female of child-bearing potential not employing adequate contraception.
13. Subjects with known hypersensitivity to peptide drugs, including LHRH agonists.
14. Receipt of 2 or more prior cytotoxic chemotherapy regimens for advanced, recurrent, or metastatic endometrial cancer.
15. Prior treatment with AEZS-108.
16. Use of LHRH agonist or antagonist treatment within 6 months prior to randomization.
17. Malignancy within last 5 years except non-melanoma skin cancer.
18. Any concomitant disease or condition which would interfere with the subjects' proper completion of the protocol assignment.
19. Concomitant or recent treatment with other investigational drug (within 4 weeks or 5 elimination half life times prior to anticipated start of study treatment).
20. Lack of ability or willingness to give informed consent.
21. Anticipated non-availability for study visits/procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Miller, MD, Principal Investigator — University of Texas Southwestern Medical Center, Dallas, USA; Hani Gabra, MD, Principal Investigator — Imperial College London Hammersmith Campus, London, UK
Locations (123):
- United States (28):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - USC Norris Hospital and LAC+USC Medical Center, Los Angeles, California
  - University of California, Irvine - Medical Center, Orange, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Women's Cancer Center, Covington, Louisiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medecine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Institute, New York, New York
  - Hope Women's Cancer Centers / Mission Hospital, Inc., Asheville, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Peggy and Charles Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - Hollings Cancer Center, MUSC, Charleston, South Carolina
  - Sanford Research/USD, Sioux Falls, South Dakota
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospitals, Falls Church, Virginia
  - Henrico Doctor's Hospital, Richmond, Virginia
  - Froedtert & The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Belarus (4):
  - Alexandrov National Cancer centre of Belarus, Minsk
  - Minsk City Clinical Oncologic Dispensary, Minsk
  - Mogilev Regional Clinical Oncologic Dispensary, Mogilev
  - Vitebsk Regional Clinical Oncologic Dispensary, Vitebsk
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - UZ Leuven - Campus Gasthuisberg, Leuven
  - Hospital Centre Liege University_CHU Sart Tilman, Liège
  - CHWAPI, Tournai
- Bosnia and Herzegovina (3):
  - Clinical Center Banja Luka, Oncology Clinic, Banja Luka
  - University Clinical Hospital Mostar, Oncology clinic, Mostar
  - Clinical Centre University of Sarajevo, Sarajevo
- Specialized Hospital for Active Treatment in Obstetrics and Gynecology, Pleven, Bulgaria
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Hopital Notre Dame - CHUM, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Hotel Dieu de Quebec- CHUQ, Québec
- Czechia (3):
  - Masarykův onkologický ústav, Brno
  - Fakultní nemocnice Olomouc, Olomouc
  - Všeobecná fakultní nemocnice v Praze, Prague
- Denmark (2):
  - Copenhagen University Hospital "Rigshospitalet", Copenhagen
  - Herlev Hospital, Herlev
- Finland (3):
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Central Hospital, Turku
- Germany (6):
  - Universitätsklinikum Köln, Cologne
  - Klinikum Frankfurt Höchst, Frankfurt
  - Georg-August-Universität Göttingen, Universitäts-Frauenklinik, Abteilung für Gynäkologie und Geburtshilfe, Göttingen
  - Universitätsklinik und Poliklinik für Gynäkologie Martin Luther Universität Halle-Wittenberg, Halle
  - University Clinic Münster, Münster
  - Klinik für Frauenheilkunde und Geburtshilfe der Universität Regensburg am Caritas-Krankenhaus St. Josef, Regensburg
- Ireland (5):
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St James's Hospital, Dublin
  - University Hospital Galway, Galway
  - Waterford Regional Hospital, Waterford
- Israel (7):
  - Barzilai Medical Center, Ashkelon
  - Rambam Health Care Campus, Haifa
  - Hadassah Hospital, Jerusalem
  - Davidoff Center, Rabin Medical Center, Petah Tikva
  - Oncology Institute Kaplan, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (6):
  - Azienda Ospedaliera Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Istituto Nazionale Tumori IRCCS, Napoli
  - Istituto Oncologico Veneto, IRCCS, Padua
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - Policlinico A. Gemelli, Rome
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Maastricht University Medical Center (UMC), Maastricht
- Norway (3):
  - Haukeland University Hospital, Bergen
  - The Norwegian Radium Hospital, Oslo
  - Helse Stavanger HF, Stavanger Universitetssjukhus, Stavanger
- Poland (5):
  - Bialostockie Centrum Onkologii, Bialystok
  - Centrum Terapii Współczesnej ul., Lodz
  - I Klinika Ginekologii Onkologicznej i Ginekologii, Lublin
  - Wojewodzki Szpital Specjalistyczny, Olsztyn
  - NZOZ Magodent, Szpital Onkologiczny, Warsaw
- Romania (6):
  - Oncolab, Craiova, Dolj
  - Spitalul Clinic Judetean Mures, Târgu Mureş, Mureș County
  - Oncology Institute "Prof. Dr. I. Chiricuta", Cluj Npaoca
  - Centru de Oncologie Sf. Nectarie, Craiova
  - Spitalul Clinic Judetean de Urgenta "Sf. Ioan cel Nou", Suceava
  - Oncomed, Timișoara
- Russia (9):
  - GAUZ "Republican Clinical Oncology Center", Kazan', Tatarstan Republic
  - FGBU "RONC n.a. N.N. Blokhin", Moscow
  - Nizhny Novgorod Regional Oncology Dispensary, Nizhny Novgorod
  - Pyatigorsk Regional Oncology Dispensary, Pyatigorsk
  - Budget Institution of Health / Leningrad Regional Oncological Dispensary, Saint Petersburg
  - Saint-Petersburg State Budgetary Institution Healthcare "City Clinical Oncology Center", Saint Petersburg
  - FGBU "NIIO n.a. N.N. Petrov", Saint Petersburg
  - Republican Clinical Oncology Dispensary, Ufa
  - Volgograd Regional Oncology Dispensary #3, Volzhskiy
- Spain (6):
  - Hospital Vall d´Hebron, Barcelona
  - MD Anderson cáncer center, Madrid
  - Ramon Y Cajal Hospital, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Instituto Valenciano de Oncologia, Valencia
- Ukraine (7):
  - Zina Memorial Cancer Hospital (LISSOD), Plyuty, Kyiv Oblast
  - Municipal institution "Dnipropetrovsk City Multidisciplinary Clinical Hospital No. 4", Dnipro
  - CCMP I Donetsk Regional Anticancer Center, Donetsk
  - Public health enterprise "Kharkov regional Clinical Oncological Center", Kharkiv
  - Kiev City Clinical Oncology Center, Kiev
  - Zakarpatskyi Regional Clinical Oncology Dispensary, Uzhhorod
  - Vinnitsa Regional Clinical Oncology Dispensary, Vinnitsa
- United Kingdom (6):
  - The Royal Marsden Hospital NHS Foundation Trust, Sutton, Surrey
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - St James's University Hospital, Leeds
  - Imperial college Healthcare NHS Trust, London
  - Nottingham City Hospital NHS Trust, Nottingham

REFERENCES:
- [Derived] Mathews C, Lorusso D, Coleman RL, Boklage S, Garside J. An Indirect Comparison of the Efficacy and Safety of Dostarlimab and Doxorubicin for the Treatment of Advanced and Recurrent Endometrial Cancer. Oncologist. 2022 Dec 9;27(12):1058-1066. doi: 10.1093/oncolo/oyac188. PMID 36124638

RESULTS

PARTICIPANT FLOW:
Groups:
- AEZS-108 / Zoptarelin Doxorubicin: 267 mg/m2 by 2-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles up to 9 cycles
  AEZS-108 / zoptarelin doxorubicin: 267 mg/m2 by 2-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles for a maximum of 9 cycles
- Doxorubicin/ Standard Chemotherapy: 60 mg/m2 by intravenous bolus injection or 1-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles
  doxorubicin: 60 mg/m2 by intravenous bolus injection or 1-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles
Period: Overall Study
Arm/Group | AEZS-108 / Zoptarelin Doxorubicin | Doxorubicin/ Standard Chemotherapy
Started (Intent-to-treat population (ITT)) | 256 (Patients allocated to AEZS-108) | 255 (Patients allocated to doxorubicin)
Modified ITT (mITT) (Excluding patients allocated to a treatment but never treated) | 252 | 249
Safety Population (SAF) | 252 | 249
Completed (Per protocol (PP) population) | 243 | 240
Not Completed | 13 | 15

BASELINE CHARACTERISTICS:
Population: ITT population, comprising all patients allocated to either AEZS-108 or doxorubicin.
Groups:
- Total: Total of all reporting groups
Arm/Group | AEZS-108 / Zoptarelin Doxorubicin | Doxorubicin/ Standard Chemotherapy | Total
Number analyzed (Participants) | 256 | 255 | 511
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 130 | 136 | 266
  >=65 years | 126 | 119 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.63) | 63.8 (8.81) | 63.7 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 256 | 255 | 511
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 237 | 240 | 477
  Race/Ethnicity: Black or African American | 10 | 7 | 17
  Race/Ethnicity: Asian | 6 | 5 | 11
  Race/Ethnicity: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Race/Ethnicity: Other | 1 | 2 | 3
  Race/Ethnicity: Unknown | 1 | 0 | 1
ECOG (Eastern Cooperative Oncology Group) PS (Performance Status) [Count of Participants; unit: Participants] — ECOG PS = Eastern Cooperation Oncology Group Performance Status.
  Status Scale Grade:
  0: Fully active, able to carry on all pre-disease Performance without restriction.
  1. Symptoms ambulatory, restricted in activity, able to carry out work of light nature
  2. In bed <50% of time, ambulatory + capable of all selfcare, unable to carry out any work activities.
  3. In bed>50% of time, capable of only limited self-care, confirmed to bed or chair >50%.
  4. 100% bedridden, completely disabled, cannot carry on any self-care. 5. Dead
  Participants
    0 | 120 | 125 | 245
    1 | 121 | 118 | 239
    2 | 15 | 11 | 26
    unknown | 0 | 1 | 1
Stage of endometrial cancer at study entry [Count of Participants; unit: Participants] — Advanced disease comprising FIGO (The International Federation of Gynecology and Obstetrics) III or IV
  Participants
    Advanced (FIGO III or IV) | 99 | 94 | 193
    Metastatic | 86 | 90 | 176
    Recurrent | 71 | 71 | 142

OUTCOME MEASURES:

1. Primary Outcome: Compare the Overall Survival (OS) of Patients Treated With AEZS-108 to the OS of Patients Treated With Doxorubicin.
Description: Overall survival was defined as the elapsed time from randomization to death from any cause. For surviving patients, follow-up was to be censored at the date of last contact.
  The final analysis, which was event-based, was conducted after approximately 384 randomized patients had died.
  A log-rank test with an overall two sided Type I Error rate of 0.05 after taking the interim analyses into account was used to compare OS between the two treatment arms via a SAS (Statistical Analysis System) LIFETEST procedure. Kaplan Meier estimates were used to calculate median OS and the 95% confidence interval (CI) of the median OS. The proportion of patients alive at 6 and 12 months (from randomization date) and the 95% CIs for these estimated proportions were calculated.
Time Frame: From randomization to death from any cause. During ongoing treatment: response evaluation every 3 cycles. For patients gone of treatment: re-assessment every 12 weeks.
Measure: Number; unit: participants
Arm/Group | AEZS-108 / Zoptarelin Doxorubicin | Doxorubicin/ Standard Chemotherapy
Number analyzed (Participants) | 256 | 255
participants
  Death Events | 196 | 188
  Censored | 60 | 67
  Survivors at 6 months | 171 | 174
  Survivors at 12 months | 111 | 106
Statistical Analysis 1: Comparison: AEZS-108 / Zoptarelin Doxorubicin; Kaplan-Meier log-log transformed estimates: survivors at 6 months; Test type: Other; Kaplan-Meier = 69.8, 95% CI 2-sided [63.6 to 75.1]
Statistical Analysis 2: Comparison: AEZS-108 / Zoptarelin Doxorubicin; Kaplan-Meier log-log transformed estimates: survivors at 12 months; Test type: Other; Kaplan-Meier = 45.8, 95% CI 2-sided [39.5 to 52.0]
Statistical Analysis 3: Comparison: Doxorubicin/ Standard Chemotherapy; Kaplan-Meier log-log transformed estimates: survivors at 6 months; Test type: Other; Kaplan-Meier = 72.1, 95% CI 2-sided [66.0 to 77.3]
Statistical Analysis 4: Comparison: Doxorubicin/ Standard Chemotherapy; Kaplan-Meier log-log transformed estimates: survivors at 12 months; Test type: Other; Kaplan-Meier = 44.6, 95% CI 2-sided [38.2 to 50.7]
Statistical Analysis 5: Comparison: AEZS-108 / Zoptarelin Doxorubicin vs Doxorubicin/ Standard Chemotherapy; A Cox model with treatment effects was used to estimate the hazard ratio and perform hypothesis testing. The estimated hazard ratio and the 95% CI of the hazard ratio were presented; Test type: Other; p = 0.5441, Log Rank; 2-sided; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.87 to 1.30]

2. Secondary Outcome: Compare Efficacy Based on Objective Response Rate (ORR).
Description: The ORR was defined as the sum of the Complete Response (CR) and Partial Response (PR).
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) was to have a reduction in the short axis to <10 mm.
  PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  All responses were confirmed at least 4 weeks after the initial response was observed. Tumor assessments occurred every 3 cycles (± 7 days) during ongoing treatment then every 3 months (± 7 days) thereafter while the patient was on study. The last assessment occurred either when progression was confirmed or when approximately 384 randomized patients had died.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | AEZS-108 / Zoptarelin Doxorubicin | Doxorubicin/ Standard Chemotherapy
Number analyzed (Participants) | 256 | 255
Participants
  CR | 6 | 5
  PR | 26 | 31
  ORR | 32 | 36
Statistical Analysis 1: Comparison: AEZS-108 / Zoptarelin Doxorubicin vs Doxorubicin/ Standard Chemotherapy; Hypothesis testing between the two treatment arms was performed using a Mantel Haenszel test. The odds ratio and 95% CI of the odds ratio were presented; Test type: Other; p = 0.5907, Mantel Haenszel; 2-sided test; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.52 to 1.45]

3. Secondary Outcome: Compare Efficacy Based on Progression-free Survival (PFS).
Description: Progression-free survival (PFS): days between randomization and the date of documented progression or death for any cause that occurred up to the end of the study. For patients whose progression status could not be determined, their PFS data was censored for the last adequate progression assessment date that the patient was confirmed to have no progression.
  Response and progression were to be evaluated using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (uni-dimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes were to be used.
  During ongoing treatment, patients were to be re-evaluated for response every 3 cycles (i.e. every 9 weeks).
  A subsequent scan was obtained no earlier than 4 weeks following the initial documentation of an objective status of either complete response (CR) or partial response (PR).
Time Frame: During ongoing treatment: response evaluation every 3 cycles. For patients gone of treatment: re-assessment every 12 weeks.
Population: The population analyzed is the mITT. PFS was analyzed in the subset of patients from mITT that have CR, PR or stable disease (SD) as best overall response.
Measure: Count of Participants; unit: Participants
Arm/Group | AEZS-108 / Zoptarelin Doxorubicin | Doxorubicin/ Standard Chemotherapy
Number analyzed (Participants) | 252 | 249
Participants
  PFS events | 166 | 148
  Censored | 90 | 107
  Progression Free Survivors at 6 months | 69 | 51
  Progression Free Survivors at 12 months | 28 | 12
Statistical Analysis 1: Comparison: AEZS-108 / Zoptarelin Doxorubicin; Kaplan-Meier log-log transformed estimates: survivors at 6 months; Test type: Other; Kaplan-Meier = 46.7, 95% CI 2-sided [39.5 to 53.6]
Statistical Analysis 2: Comparison: AEZS-108 / Zoptarelin Doxorubicin; Kaplan-Meier log-log transformed estimates: survivors at 12 months; Test type: Other; Kaplan-Meier = 20.6, 95% CI 2-sided [14.6 to 27.4]
Statistical Analysis 3: Comparison: Doxorubicin/ Standard Chemotherapy; Kaplan-Meier log-log transformed estimates: survivors at 6 months; Test type: Other; Kaplan-Meier = 47.5, 95% CI 2-sided [40.0 to 54.7]
Statistical Analysis 4: Comparison: Doxorubicin/ Standard Chemotherapy; Kaplan-Meier log-log transformed estimates: survivors at 12 months; Test type: Other; Kaplan-Meier = 12.3, 95% CI 2-sided [6.9 to 19.3]
Statistical Analysis 5: Comparison: AEZS-108 / Zoptarelin Doxorubicin vs Doxorubicin/ Standard Chemotherapy; Hypothesis testing between the two treatment arms was performed using a log rank test; Test type: Other; p = 0.3089, Log Rank; 2-sided; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.71 to 1.11]

4. Secondary Outcome: Compare Efficacy Based on Clinical Benefit Rate (CBR).
Description: Clinical benefit was defined as having stable disease (SD) or better lasting for at least 9 weeks. The CBR was analyzed using the same methods for the ORR analyses. The analysis of CBR (CR+PR+SD) was performed in the ITT (intention-to-treat) population.
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) was to have a reduction in the short axis to <10 mm.
  PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  All responses were confirmed at least 4 weeks after the initial response was observed. Tumor assessments occurred every 3 cycles (± 7 days) during ongoing treatment then every 3 months (± 7 days) thereafter while the patient was on study. The last assessment occurred either when progression was confirmed or when approximately 384 randomized patients had died.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | AEZS-108 / Zoptarelin Doxorubicin | Doxorubicin/ Standard Chemotherapy
Number analyzed (Participants) | 256 | 255
Participants
  CR | 6 | 5
  PR | 26 | 31
  SD | 106 | 102
  Progressive Disease (PD) | 65 | 67
Statistical Analysis 1: Comparison: AEZS-108 / Zoptarelin Doxorubicin vs Doxorubicin/ Standard Chemotherapy; Hypothesis testing between the two treatment arms was performed using a Mantel Haenszel test; Test type: Other; p = 0.6924, Mantel Haenszel; 2-sided; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.76 to 1.52]

ADVERSE EVENTS:
Time Frame: Approx. over 3 years, during the whole duration of the trial.
Description: The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; version 4.03 or subsequent ones) were to be used for the grading of severity of symptoms and abnormal findings.
Groups:
- AEZS-108 / Zoptarelin Doxorubicin: 267 mg/m^2 by 2-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles up to 9 cycles
  AEZS-108 / zoptarelin doxorubicin: 267 mg/m2 by 2-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles for a maximum of 9 cycles
- Doxorubicin/ Standard Chemotherapy: 60 mg/m^2 by intravenous bolus injection or 1-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles
  doxorubicin: 60 mg/m2 by intravenous bolus injection or 1-hour intravenous infusion, on Day 1 of 21-day (3-week) cycles
Arm/Group | AEZS-108 / Zoptarelin Doxorubicin | Doxorubicin/ Standard Chemotherapy
All-Cause Mortality (participants affected / at risk) | 196/252 | 188/249
Serious Adverse Events (participants affected / at risk) | 92/252 | 75/249
Other Adverse Events (participants affected / at risk) | 239/252 | 240/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AEZS-108 / Zoptarelin Doxorubicin (N=252) | Doxorubicin/ Standard Chemotherapy (N=249)
Neutropenia (Blood and lymphatic system disorders) | 21 | 15
Anemia (Blood and lymphatic system disorders) | 16 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 17 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 3
Nause (Gastrointestinal disorders) | 11 | 8
Vomiting (Gastrointestinal disorders) | 7 | 9
Leukopenia (Blood and lymphatic system disorders) | 4 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dehydratation (Metabolism and nutrition disorders) | 8 | 2
Dyspnoe (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Intestinal obstruction (Gastrointestinal disorders) | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AEZS-108 / Zoptarelin Doxorubicin (N=252) | Doxorubicin/ Standard Chemotherapy (N=249)
Neutropenia (Blood and lymphatic system disorders) | 132 | 126
Nausea (Gastrointestinal disorders) | 120 | 125
Aneamia (Blood and lymphatic system disorders) | 107 | 101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
According to the study protocol, "draft versions of abstracts or manuscripts must be made available to the co-authors and to the sponsor before any presentation of results or submission for publication. At least 3 weeks should be allowed for review and comment of an abstract and 4 weeks in case of a full paper, respectively. Multiple review cycles are usual for full papers and respective planning must account for this." In addition, the definitions per individual trial site agreement did apply.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT01767155/SAP_000.pdf
  • Study Protocol (2014-09-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT01767155/Prot_001.pdf